CLINICAL TRIAL: NCT02318355
Title: Resuscitative Effect of Two Liters of Crystalloid on Hemodilution and Base Deficit in Healthy Volunteer Blood Donors With Class I Hemorrhage.
Brief Title: Proving Hemodilution in a Human Model for Class I Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Community Blood Center of the Carolinas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-08-19E
Record Dates: First submitted 2014-12-10; First posted 2014-12-17 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2014-12

CONDITIONS: Hemodilution; Hemorrhage; Shock; Wounds and Injuries
Keywords: hemodilution; hemorrhage; trauma; lactate; base deficit; randomized control trial
MeSH Terms: conditions — Hemorrhage; Shock; Wounds and Injuries | interventions — Saline Solution; Ringer's Lactate

ARMS (3):
- Control (No Intervention): Control group that receives no intravenous fluid after blood donation
- Lactated Ringers (Experimental): Experimental group that receives two liters lactated ringers after blood donation.
  Interventions: Other: lactated ringers
- Normal Saline (Experimental): Experimental group that receives two liters normal saline after blood donation.
  Interventions: Other: normal saline

INTERVENTIONS:
Other: normal saline — Crystalloid intravenous solution
  Other Names: NS
  Arms: Normal Saline
Other: lactated ringers — Crystalloid intravenous solution
  Other Names: LR
  Arms: Lactated Ringers

SUMMARY:
This study is a randomized control trial in volunteer blood donors to quantify the effect of blood loss and subsequent crystalloid infusion on hemoglobin and markers of resuscitation such as base deficit and lactate.

DETAILED DESCRIPTION:
Blood donors were randomized to one of three arms after donation of 500cc of blood. The control group received no intravenous fluids, while donors in the two intervention arms wither received two liters normal saline or lactated ringers. Chemistries and blood gases were obtained before donation, after donation and after resuscitation. Donors hemoglobin levels were then compared over time and between study arms. Additionally, lactate and base deficit, which are markers of shock, will be collected at the time points as well to measure their response to resuscitation. Standard statistical tests were used to compare the laboratory values between groups.

ELIGIBILITY:
Inclusion Criteria:

* blood bank inclusion criteria for donation
* able to donate 500cc blood
* age > or = 18

Exclusion Criteria:

* unable to obtain IV access
* multiple blood draws fail to run on laboratory assays

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (g/dL) | 2 hours
  obtain hemoglobin immediately before and after donation, and after resuscitation with intravenous fluids. From donation to end of resuscitation, the time frame will be 2 hours or less. Donors will not be followed after the third blood draw and will be discharged from the study. No follow-up was obtained.

SECONDARY OUTCOMES:
Lactate (mmol/L) | 2 hours
  Obtain lactate immediately before and after donation, and after resuscitation with intravenous fluids. Lactate is a measure of aneorbic metabolism and increases with worsening shock and hypoperfusion as seen in hemorrhage. From donation to end of resuscitation, the time frame will be 2 hours or less. Donors will not be followed after the third blood draw and will be discharged from the study. No follow-up was obtained.
Base deficit (mmol/L) | 2 hours
  Obtain base deficit immediately before and after donation, and after resuscitation with intravenous fluids. Base deficit is a measure of unmeasured acid in the blood, indicating acidosis and shock, and increases in worsening hypoperfusion. From donation to end of resuscitation, the time frame will be 2 hours or less. Donors will not be followed after the third blood draw and will be discharged from the study. No follow-up was obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald F Sing, DO, Principal Investigator — Professor of Surgery

REFERENCES:
- [Derived] Ross SW, Christmas AB, Fischer PE, Holway H, Seymour R, Huntington CR, Heniford BT, Sing RF. Defining Dogma: Quantifying Crystalloid Hemodilution in a Prospective Randomized Control Trial with Blood Donation as a Model for Hemorrhage. J Am Coll Surg. 2018 Sep;227(3):321-331. doi: 10.1016/j.jamcollsurg.2018.05.005. Epub 2018 Jun 4. PMID 29879520
- [Derived] Ross SW, Christmas AB, Fischer PE, Holway H, Walters AL, Seymour R, Gibbs MA, Heniford BT, Sing RF. Impact of common crystalloid solutions on resuscitation markers following Class I hemorrhage: A randomized control trial. J Trauma Acute Care Surg. 2015 Nov;79(5):732-40. doi: 10.1097/TA.0000000000000833. PMID 26496098